CLINICAL TRIAL: NCT04588103
Title: The Effects of 8 Weeks of Lower Limb Heat Therapy, Moderate-intensity Cycling Exercise, or Both on Vascular Function in Young, Healthy Males and Females
Brief Title: Artery Function Responses to Heat Therapy and Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HEATEX
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Endothelial Dysfunction
Keywords: heat therapy; exercise training; endothelial function
MeSH Terms: conditions — Hyperthermia | interventions — Diathermy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will be asked to maintain their regular physical activity habits for the duration of the 8-week intervention period.
- Heat therapy (Experimental): Participants will be asked to undergo 45 minutes of lower limb hot water immersion (42 degrees C) 3 times per week for 8 weeks.
  Interventions: Other: Heat therapy
- Exercise training (Experimental): Participants will be asked to undergo 45 minutes of moderate-intensity cycling exercise (~40-59% VO2 reserve) 3 times per week for 8 weeks.
  Interventions: Other: Exercise training
- Combined training (Experimental): Participants will be asked to undergo 90 minutes of moderate-intensity cycling exercise and lower limb hot water immersion sequentially 3 times per week for 8 weeks.
  Interventions: Other: Heat therapy; Other: Exercise training

INTERVENTIONS:
Other: Heat therapy — Lower limb warm water immersion (42 degrees C)
  Arms: Combined training; Heat therapy
Other: Exercise training — Moderate-intensity cycling exercise (~40-59% VO2 reserve)
  Arms: Combined training; Exercise training

SUMMARY:
This study will explore the effects of 8 weeks of local leg heat therapy, exercise training, or both on measures of vascular function, cardiorespiratory fitness, and muscle strength in young, healthy individuals. Participants will be allocated into either a control group that will maintain their regular physical activity habits; or into one of three training groups: heat therapy will involve lower limb warm water immersion, exercise training will involve moderate-intensity cycling, and combined training will involve both performed in sequential order.

DETAILED DESCRIPTION:
A between-groups interventional design will be used in a cohort of 80 young, healthy males and females 18-35 years old. Interested individuals will be invited to the lab for a screening and familiarization visit (1 hr), in which participants will be introduced to various lab testing protocols to ensure proper performance and tolerance during experimental data collection sessions. Participants will be randomized into one of four groups for an 8-week intervention period: (1) no training (CON), (2) lower limb heat therapy (HEAT), (3) moderate intensity cycling training (EX), or (4) combined training (HEATEX). CON will involve maintenance of regular physical activity habits. HEAT will involve 45 minutes of lower limb hot water immersion (42 °C) using a custom-made heating apparatus 3x/week. EX will involve of 45 minutes of cycling on an ergometer at 40-59% VO2reserve 3x/week. HEATEX will require participants to perform 3x/week of exercise training and heat therapy consecutively and in that order, such that each session is 90 minutes in duration. In total, all groups except CON will be expected to complete 24 intervention sessions. Vascular function will be characterized by measures of endothelial function, arterial stiffness, arterial structure, central hemodynamics, arterial blood flow and shear, and endothelial cell nitric oxide production. Muscle and metabolic adaptations will be characterized by measures of cardiorespiratory fitness, body composition, muscle strength and thickness, and fasting glucose and insulin. Inflammatory profile will be characterized by concentrations of interleukins, heat shock proteins, and cortisol. Thermal physiological adaptations will be characterized by measures of core and skin temperature and sweat rate. Perceptual responses will be characterized by measures of thermal comfort and sensation, calmness, alertness, mood, affect, and ratings of perceived exertion. Intervention adherence will be tracked throughout the intervention period. For the acute investigation (3-hr visit), outcome measures will be assessed before and immediately following the first and last training session. For the chronic investigation (2-hr visit), outcome measures will be assessed at weeks 0, 2, 4, 6, and 8 of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (i.e., no cardiovascular, musculoskeletal, or metabolic disease)
* 18-35 years old
* Recreationally and/or physically active

Exclusion Criteria:

* History of cardiovascular, musculoskeletal, or metabolic disease
* Regular smoking and/or vasoactive drug use

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Brachial artery endothelial function | Change in endothelial function from week 0 to 8
  Flow-mediated dilation (FMD) is a measure of the ability of the artery to dilate in response to elevated shear stress, and represents endothelial function. For this technique, a pressure cuff will be wrapped around the forearm and then inflated to ~200 mmHg for 5 minutes to occlude blood flow through the artery site. Doppler ultrasound (Vivid q, GE Medical Systems, Horten, Norway) and a 12 MHz linear array probe will be used to measure artery diameter before cuff inflation (rest), before cuff deflation (ischemia), and for three minutes after cuff deflation (reactive hyperemia). Images of the BA will be collected in Duplex mode and obtained proximal to the antecubital fossa. FMD will be calculated using this formula: FMD% = ((peak diameter-baseline diameter)/baseline diameter) × 100%.
Arterial stiffness | Change in arterial stiffness from week 0 to 8
  Pulse wave velocity (PWV) is a measure of the speed at which a pulse travels between two superficial artery sites, and represents arterial stiffness. For this outcome, applanation tonometers (i.e., micromanometer-tipped probes) (SPT-301, Millar Instruments, Houston, Texas, USA) will be used to detect and transmit pulse pressure wave forms at the carotid, femoral, and dorsalis pedis or tibialis posterior arteries. PWV will be calculated between the carotid-femoral arteries and femoral-foot arteries to quantify central and peripheral arterial stiffness, respectively, using this general formula: PWV = distance/pulse transit time.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Change in cardiorespiratory fitness from week 0 to 8
  VO2peak represents the maximum rate of oxygen consumption that the body can attain, and is reliant on both oxygen delivery to muscles and oxygen utilization by muscles. In this VO2peak test, participants will cycle on a cycle ergometer (Excalibur Lode B.V., Groningen, The Netherlands) at an intensity that begins at 50 W and progressively increases at a rate of 1 W every 2 seconds until volitional exhaustion or a pedaling cadence < 60 rpm. A mask equipped with a breath-by-breath gas analyzer (Quark CPET, COSMED, Rome, Italy) will be worn to obtain the ratio of CO2 produced to O2 consumed, and a HR monitor (Polar Electro Oy, Kempele, Finland) will be worn to monitor HR throughout the duration of the test. VO2peak will be calculated using this formula: VO2peak = (VI * FIO2) - (VE * FEO2).
Body composition | Change in body composition from week 0 to 8
  Body composition tests measure the proportions of fat mass and fat-free mass in the body. Participants will have their body composition assessed through air displacement plethysmography (BodPod). This method is non-invasive and involves ~5 minutes of sitting still and quietly as the measurement is completed.
Muscle strength | Change in muscle strength from week 0 to 8
  Knee extensor muscle strength will be assessed with an isokinetic dynamometer (Biodex). Participants will be familiarized with the testing procedures before assessment. Participants will be seated with restraining straps secured over the trunk, pelvis, and thigh; arms will be crossed over their chest. The axis of the dynamometer will be aligned with the axis of rotation of the knee joint. Participants will be asked to kick out repeatedly against the arm of the machine, and the force produced will be recorded.
Metabolic blood markers | Change in metabolic markers from week 0 to 8
  Fasting insulin and glucose will be measured in blood plasma and serum.
Core temperature | Change in core temperature from week 0 to 8
  Core temperature will be measured using a wireless telemetric pill during the acute experimental testing visits, and tympanic and rectal thermometry during all experimental testing visits. Participants will be instructed to swallow the pill with water 2-3 hours prior to each testing session.
Endothelial cell nitric oxide production markers | Change in endothelial nitric oxide production from week 0 to 8
  Endothelial nitric oxide synthase protein content and activity, and nitric oxide and superoxide anion production will be measured in human umbilical vein endothelial cell cultures bathed in serum collected from the study.
Heat shock protein mRNA and content | Change in heat shock proteins from week 0 to 8
  HSP72 and HSP90 will be measured in blood plasma and serum.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen J MacDonald, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Vascular Dynamics Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng JL, MacDonald MJ. Effect of heat stress on vascular outcomes in humans. J Appl Physiol (1985). 2019 Mar 1;126(3):771-781. doi: 10.1152/japplphysiol.00682.2018. Epub 2019 Jan 24. PMID 30676869
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Gimbrone MA Jr, Garcia-Cardena G. Endothelial Cell Dysfunction and the Pathobiology of Atherosclerosis. Circ Res. 2016 Feb 19;118(4):620-36. doi: 10.1161/CIRCRESAHA.115.306301. PMID 26892962
- [Background] Heinonen I, Laukkanen JA. Effects of heat and cold on health, with special reference to Finnish sauna bathing. Am J Physiol Regul Integr Comp Physiol. 2018 May 1;314(5):R629-R638. doi: 10.1152/ajpregu.00115.2017. Epub 2017 Dec 20. PMID 29351426
- [Background] Miyata M, Tei C. Waon therapy for cardiovascular disease: innovative therapy for the 21st century. Circ J. 2010 Apr;74(4):617-21. doi: 10.1253/circj.cj-09-0939. Epub 2010 Feb 13. PMID 20154403
- [Background] Serbulea M, Payyappallimana U. Onsen (hot springs) in Japan--transforming terrain into healing landscapes. Health Place. 2012 Nov;18(6):1366-73. doi: 10.1016/j.healthplace.2012.06.020. Epub 2012 Jul 17. PMID 22878276
- [Background] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Background] Van Bortel LM, Laurent S, Boutouyrie P, Chowienczyk P, Cruickshank JK, De Backer T, Filipovsky J, Huybrechts S, Mattace-Raso FU, Protogerou AD, Schillaci G, Segers P, Vermeersch S, Weber T; Artery Society; European Society of Hypertension Working Group on Vascular Structure and Function; European Network for Noninvasive Investigation of Large Arteries. Expert consensus document on the measurement of aortic stiffness in daily practice using carotid-femoral pulse wave velocity. J Hypertens. 2012 Mar;30(3):445-8. doi: 10.1097/HJH.0b013e32834fa8b0. PMID 22278144
- [Result] Bailey TG, Cable NT, Miller GD, Sprung VS, Low DA, Jones H. Repeated Warm Water Immersion Induces Similar Cerebrovascular Adaptations to 8 Weeks of Moderate-Intensity Exercise Training in Females. Int J Sports Med. 2016 Sep;37(10):757-65. doi: 10.1055/s-0042-106899. Epub 2016 Jun 10. PMID 27286178
- [Result] Brunt VE, Eymann TM, Francisco MA, Howard MJ, Minson CT. Passive heat therapy improves cutaneous microvascular function in sedentary humans via improved nitric oxide-dependent dilation. J Appl Physiol (1985). 2016 Sep 1;121(3):716-23. doi: 10.1152/japplphysiol.00424.2016. Epub 2016 Jul 14. PMID 27418688
- [Result] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Result] Carter HH, Spence AL, Atkinson CL, Pugh CJ, Naylor LH, Green DJ. Repeated core temperature elevation induces conduit artery adaptation in humans. Eur J Appl Physiol. 2014 Apr;114(4):859-65. doi: 10.1007/s00421-013-2817-2. Epub 2014 Jan 8. PMID 24399113
- [Result] Gurovich AN, Braith RW. Enhanced external counterpulsation creates acute blood flow patterns responsible for improved flow-mediated dilation in humans. Hypertens Res. 2013 Apr;36(4):297-305. doi: 10.1038/hr.2012.169. Epub 2012 Oct 18. PMID 23076403
- [Result] Hesketh K, Shepherd SO, Strauss JA, Low DA, Cooper RJ, Wagenmakers AJM, Cocks M. Passive heat therapy in sedentary humans increases skeletal muscle capillarization and eNOS content but not mitochondrial density or GLUT4 content. Am J Physiol Heart Circ Physiol. 2019 Jul 1;317(1):H114-H123. doi: 10.1152/ajpheart.00816.2018. Epub 2019 May 10. PMID 31074654
- [Result] Hoekstra SP, Bishop NC, Faulkner SH, Bailey SJ, Leicht CA. Acute and chronic effects of hot water immersion on inflammation and metabolism in sedentary, overweight adults. J Appl Physiol (1985). 2018 Dec 1;125(6):2008-2018. doi: 10.1152/japplphysiol.00407.2018. Epub 2018 Oct 18. PMID 30335579
- [Result] Hunter SD, Dhindsa MS, Cunningham E, Tarumi T, Alkatan M, Nualnim N, Elmenshawy A, Tanaka H. The effect of Bikram yoga on endothelial function in young and middle-aged and older adults. J Bodyw Mov Ther. 2017 Jan;21(1):30-34. doi: 10.1016/j.jbmt.2016.06.004. Epub 2016 Jun 17. PMID 28167186
- [Result] Jakubowski JS, Wong EPT, Nunes EA, Noguchi KS, Vandeweerd JK, Murphy KT, Morton RW, McGlory C, Phillips SM. Equivalent Hypertrophy and Strength Gains in beta-Hydroxy-beta-Methylbutyrate- or Leucine-supplemented Men. Med Sci Sports Exerc. 2019 Jan;51(1):65-74. doi: 10.1249/MSS.0000000000001752. PMID 30113522
- [Result] Schlader ZJ, Gagnon D, Adams A, Rivas E, Cullum CM, Crandall CG. Cognitive and perceptual responses during passive heat stress in younger and older adults. Am J Physiol Regul Integr Comp Physiol. 2015 May 15;308(10):R847-54. doi: 10.1152/ajpregu.00010.2015. Epub 2015 Mar 18. PMID 25786484
- [Result] Totosy de Zepetnek JO, Ditor DS, Au JS, MacDonald MJ. Impact of shear rate pattern on upper and lower limb conduit artery endothelial function in both spinal cord-injured and able-bodied men. Exp Physiol. 2015 Oct;100(10):1107-17. doi: 10.1113/EP085056. Epub 2015 Aug 18. PMID 26206681
- [Derived] Cheng JL, Pizzola CA, Mattook KC, Noguchi KS, Armstrong CM, Bagri GK, Macdonald MJ. Effects of Lower Limb Heat Therapy, Exercise Training, or a Combined Intervention on Vascular Function: A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Jan 1;57(1):94-105. doi: 10.1249/MSS.0000000000003550. Epub 2024 Sep 16. PMID 39283227